CLINICAL TRIAL: NCT02332967
Title: Safety and Efficacy of Addition of Structured Lipids in Starter Formulas
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Société des Produits Nestlé (SPN) (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 06.16.INF
Record Dates: First submitted 2014-10-30; First posted 2015-01-07 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2014-11

CONDITIONS: Healthy Newborn Infants
MeSH Terms: interventions — Palmitic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Whey predominant starter formula (Active Comparator): Whey predominant starter formula
  Interventions: Other: Whey predominant starter formula + 40% palmitic acid; Other: Whey predominant starter formula + 50% palmitic acid
- Whey predominant starter formula + 40% palmitic acid (Experimental): Whey predominant starter formula + 40% palmitic acid in sn-2 position
  Interventions: Other: Whey predominant starter formula
- Whey predominant starter formula + 50% palmitic acid (Experimental): Whey predominant starter formula + 50% palmitic acid in sn-2 position
  Interventions: Other: Whey predominant starter formula

INTERVENTIONS:
Other: Whey predominant starter formula — Milk powder product given to babies between 1 week and 4 months
  Arms: Whey predominant starter formula + 40% palmitic acid; Whey predominant starter formula + 50% palmitic acid
Other: Whey predominant starter formula + 40% palmitic acid — Milk powder product containing 40% of palmitic acid
  Arms: Whey predominant starter formula
Other: Whey predominant starter formula + 50% palmitic acid — Milk powder product containing 50% of palmitic acid
  Arms: Whey predominant starter formula

SUMMARY:
The primary objective of this trial is to demonstrate that infants receiving an infant formula in which 40 or 50% of the palmitic acid is in the sn-2 position have, during the first 4 months of life, stools that are softer than those of infants receiving a control formula.

DETAILED DESCRIPTION:
Human milk is considered as the golden standard for infant formula. In human milk and infant formula lipids provide about 55% of energy for the infant and represent as such a major nutrient for the baby. The vast majority of the lipids in human milk is composed of triacylglycerols (98% of total lipids) and the remainder percent are phospholipids. Triglycerides are composed of the glycerol backbone to which three fatty acids are bound. In human milk, palmitate (16:0) is the major long chain saturated fatty acid representing 22% to 26% of total fatty acids, esterified to approximately 70% in sn-2 position on the glycerol backbone. Unsaturated fatty acids such as oleic acid (18:1) and linoleic acid (18:2n-6) are preferentially esterified at the 1 and 3 position. In infant formulas the major source of palmitic acid is palm oil or palm olein where palmitate is, however, preferentially in the external 1,3 positions, and mono- and polyunsaturated fatty acids are usually esterified at the 2-position of the triacylgycerol.

The aim of this study is to assess the safety and efficacy of infant formula containing 40% and 50%, respectively, of palmitic acid in sn-2 position.

ELIGIBILITY:
Inclusion Criteria:

* healthy newborn infants
* full term infant (37 - 42 weeks gestation)
* birth weight between 2.5 and 4.5 kg
* singleton birth
* the infant's mother has elected to exclusively formula feed her baby, from enrollment to 4 months of age
* having obtained his7her legal representative's informed consent

Exclusion Criteria:

* congenital illness or malformation that may affect normal growth
* significant pre-natal and/or post-natal disease
* hospitalization in the first 14 days of life after the child has left the maternity ward
* receiving antibiotic treatment at time of enrolment
* newborn whose parents/caregivers cannot be expected to comply with treatment
* newborn currently participating in another interventional clinical trial.

Ages: 1 Week to 4 Months | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 488 (Actual)
Dates: Start 2007-07; Primary Completion 2012-02 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Stool consistency | 4 months
  To demonstrate that the infants receiving an infant formula with 40% or 50% of palmitic acid during the first 4 months of life have softer stools than the ones receiving the control formula.
Baby weight gain | 4 months
  To demonstrate that the weight gain in babies receiving the experimental formula is the same as with the control formula

SECONDARY OUTCOMES:
Baby length and head circumference | 4 months
  To assess whether the groups have comparable changes in length, and head circumference
Digestive tolerance using a questionnaire filled in by the mothers | 4 months
  To assess the infants' digestive tolerance of the starter formula
Gut microbiota using microbiology method | 4 months
  To compare gut microbiota between the groups
Fat quantity in the stools | 4 months
  To assess fat absorption
Baby body composition (DEXA) | 4 months
  To compare body composition
Food intake by the baby | 4 months
  To compare volume intake between the groups
Rate of spitting up | 4 months
  To compare spitting up between the groups
Number of adverse events | 4 months
  To evaluate the frequency of episodes of morbidity (adverse events)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique Turck, Prof, Principal Investigator — Gatroenterology and Nutrition, Pediatric dept, CHRU Lille

REFERENCES:
- [Derived] Beghin L, Marchandise X, Lien E, Bricout M, Bernet JP, Lienhardt JF, Jeannerot F, Menet V, Requillart JC, Marx J, De Groot N, Jaeger J, Steenhout P, Turck D. Growth, stool consistency and bone mineral content in healthy term infants fed sn-2-palmitate-enriched starter infant formula: A randomized, double-blind, multicentre clinical trial. Clin Nutr. 2019 Jun;38(3):1023-1030. doi: 10.1016/j.clnu.2018.05.015. Epub 2018 Jun 1. PMID 29903473